CLINICAL TRIAL: NCT03189316
Title: Can the Peritoneal Cavity be a Source of Regulatory B Cells to Treat Auto-immune Disease?
Brief Title: Anti-inflammatory Cells in Peritoneal Cavity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Absence of BReg Lymphocytes in peritoneum
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 9828
Record Dates: First submitted 2017-05-30; First posted 2017-06-16 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Ovarian Cysts; Chronic Renal Insufficiency
Keywords: Peritoneal fluid; B cells; Regulatory B cells; Human
MeSH Terms: conditions — Ovarian Cysts; Renal Insufficiency, Chronic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- subjects with ovarian cyst (Other): Peritoneal fluid sample obtained from coelioscopy for exploration of ovarian cysts and blood sample
  Interventions: Other: peritoneal fluid and blood sample
- subjects with peritoneal dialysis (Other): Peritoneal fluid sample obtained from peritoneal dialysis fluid of patients with chronic renal insufficiency and blood sample
  Interventions: Other: peritoneal fluid and blood sample

INTERVENTIONS:
Other: peritoneal fluid and blood sample — Peritoneal fluid sample obtained from peritoneal dialysis fluid of patients with chronic renal insufficiency and blood sample or Peritoneal fluid obtained from coelioscopy for exploration of ovarian cysts and blood cell

SUMMARY:
Some subsets of lymphocytes are able to inhibit immune response and thus, could be used to control auto-immune diseases and transplant reject. In mice, the main source of those anti-inflammatory lymphocytes is the peritoneal cavity. No data are available in human. This study aims at exploring the presence of those anti-inflammatory lymphocytes in human peritoneal cavity and at determine how to expand those cells.

DETAILED DESCRIPTION:
B cells will be collected during procedures planned for patients' standard care. Peritoneal fluid and peripheral blood of patients will be collected during coelioscopy for exploration of ovarian cysts or dialysis for treatment of chronic renal insufficiency.

Regulatory B cells (Breg cells) will be measured in peritoneal fluid and in peripheral blood after in vitro stimulation and assessment of intracellular interleukin-10 by flow cytometry. Proportion of Breg cells among B cells will be compared between peritoneal fluid and peripheral blood in both groups.

Different protocols to induce differentiation of B cells into Breg cells will be tested and compared.

ELIGIBILITY:
Inclusion criteria:

* woman over 18 year old undergoing exploration of ovarian cysts by coelioscopy
* patient with chronic renal insufficiency undergoing peritoneal dialysis
* informed consent obtained

Exclusion criteria:

* pregnancy or breast-feeding
* non affiliation to health care insurance
* treatment with corticosteroids over 15 mg/day
* treatment with rituximab

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-13 (Actual)

PRIMARY OUTCOMES:
relative percentage of regulatory B cells among B cells in peritoneal cavity compared to peripheral blood | up to 48 hour
  Comparison of Breg cell in peritoneal cavity to Breg cell in peripheral blood B

CONTACTS AND LOCATIONS:
Locations (1):
- CHU montpellier - department of rheumatology, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided